CLINICAL TRIAL: NCT06208345
Title: Early Life Intervention in Pediatrics Supported by E-health (ELIPSE I): Coaching Parents to Lower Obesity in Children. A Single-blind Randomized Controlled Parallel-group Clinical Trial.
Brief Title: Early Life Intervention in Pediatrics Supported by E-health
Acronym: ELIPSE-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5519; 2023-01136 (Other: KEK Bern)
Record Dates: First submitted 2023-12-19; First posted 2024-01-17 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Adiposity; Childhood Obesity; Adolescent Obesity; Non-communicable Disease; Life Style; Behavior, Eating; Behavior, Health
Keywords: Adiposity; Children; Adolescents; Prevention; eHealth
MeSH Terms: conditions — Obesity; Pediatric Obesity; Noncommunicable Diseases; Feeding Behavior; Health Behavior

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled parallel-group clinical trial
Who Masked: Care Provider, Investigator
Masking Description: The treating physicians are kept blind to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) with Life-Style app (Experimental): Children in the intervention group receive treatment as usual (TAU) and the parents receive a smartphone app during the main intervention period of 20 weeks. The app (life-style app) aims to promote healthy behaviour through cognitive-behavioural impact factors.
  Interventions: Behavioral: Life-Style app
- Treatment as usual (TAU) (No Intervention): The children in the control group only receive treatment-as-usual (TAU) and the parents do not have an active app during the main intervention period of 20 weeks. TAU includes lifestyle behaviour counselling, dietary counselling by specialized dieticians, prescriptions for physiotherapy, as provided at the last clinical visit.

INTERVENTIONS:
Behavioral: Life-Style app — The modules of the Life-Style app are introduced and unlocked sequentially during the first weeks of the intervention phase. Afterwards the modules are fully available. Duration and frequency of app-use is not limited. The parents are accompanied by a coach through the app, who gives regular structured feedback and individual inputs. The coach has access to all data collected in the app.
  Other Names: Smartphone App
  Arms: Treatment as usual (TAU) with Life-Style app

SUMMARY:
Childhood obesity in early life contributes to the development of specific NCDs, i.e. adult obesity. Unhealthy diet and low level of physical activity are lifestyle risk behaviors associated with chronic, systemic inflammation, which promotes the pathogenesis of NCDs. Early preventive measures to improve lifestyle behavior are of utmost importance. The aim of ELIPSE-I is to assess whether an eHealth application intervention for parents is feasible and efficacious in lowering total energy intake/total energy expenditure (TEI/TEE) ratio in their children with BMI >97 centile (ELIPSE-I).

DETAILED DESCRIPTION:
ELIPSE-I represents a single-blind randomized controlled parallel-group clinical trial. In ELIPSE-I, 148 children, matched for sex, 6-12 years of age with a BMI >97 centile based on national growth charts will be included. Children will be recruited at the children's university hospital and randomly (1:1) assigned to a control and intervention group. All participants receive treatment-as-usual (TAU), parents of participants in the intervention group additionally receive a smartphone application (lifestyle app) for 20 weeks. The app aims to promote healthy behavior through cognitive-behavioral impact factors (i.e., psychoeducation, goal setting), that are applied by a psychologist via structured feedback. Single-blinded assessments will be conducted at baseline, following the intervention period of 20 weeks, and at 6-month follow-up after the end of the intervention. The primary endpoint is reduction of the TEI/TEE ratio in children with obesity. Secondary endpoints in ELIPSE-I include lowering the severity of obesity, cardiometabolic risk factor improvement, reduction in chronic low-level inflammatory biomarkers, and improved children's quality of life. A further endpoint is acceptance and usability of the app.

ELIGIBILITY:
Inclusion Criteria:

* German speaking parents
* Any ethnic background/race
* Children should live/grow-up in the same household as the parental participant
* Children with an age- and sex-matched BMI >97 centile according to Swiss national growth charts
* Children who newly attend the outpatient weight management clinic at the Division of Pediatric Endocrinology at the University Children's Hospital Bern
* Signed informed consent form from parent(s)

Exclusion Criteria:

* Syndromic obesity
* Known congenital disease affecting musculo-skeletal, cardiac or pulmonary function
* Participation in another clinical trial targeting similar objectives

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in TEI/TEE ratio | +22 weeks (Post intervention)
  TEI will be assessed by trained paediatric dietitians collecting 24-h dietary recalls on 3 days at baseline, post intervention and follow-up. TEE will be calculated using bio-impedance related body composition measures according to formulas provided by Pontzer et al. (2021; PMID: 34385400)
Change from baseline in TEI/TEE ratio | +48 weeks (Follow-Up)
  TEI will be assessed by trained paediatric dietitians collecting 24-h dietary recalls on 3 days at baseline, post intervention and follow-up. TEE will be calculated using bio-impedance related body composition measures according to formulas provided by Pontzer et al. (2021; PMID: 34385400)

SECONDARY OUTCOMES:
Change in BMI z-score | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  BMI z-score will be calculated from height and weight data, considering age and sex, according to national and international representative growth charts
Change in %>95th BMI-centile | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  The %>95th BMI-centile is a continuous measure starting from the 95th BMI-centile, and is a ratio of the individual's BMI divided by the relevant 95th BMI-centile for an age- and sex-matched individual multiplied by 100 %
Change in body fat percentage | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  The % bodyfat will be measured with a four-point bio-impedance device
Change in waist circumference | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  The waist circumference will be measured midway between iliac crest and lower end of ribs to the nearest 0.5 cm with a non-stretchable meter
Cardiometabolic risk factor response: Change in 24-hours ambulatory blood pressure | Baseline, +22 weeks (Post intervention)
  24-hours ambulatory blood pressure measurements (ABPM) are assessed at baseline and post intervention.
Cardiometabolic risk factor response: Change in carotid-femoral pulse wave velocity | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Carotid-femoral pulse wave velocity (PWV) to assess arterial stiffness
Cardiometabolic risk factor response: Change in plasma glucose levels | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Fasting plasma glucose levels are assessed for detection of insulin resistance
Cardiometabolic risk factor response: Change in lipid levels | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Fasting lipid profiles are assessed
Cardiometabolic risk factor response: Change in insulin levels | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Fasting insulin levels are measured for detection of insulin resistance
Cardiometabolic risk factor response: Change in HbA1c levels | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  HbA1c levels are assessed
Chronic low-level inflammatory biomarkers: Change in white blood cell count | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  White blood cell count as inflammatory biomarker to assess chronic low-level inflammation.
Chronic low-level inflammatory biomarkers: Change in high-sensitivity C-reactive protein (hs-CRP) | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  High-sensitivity C-reactive protein (hs-CRP) as inflammatory biomarker to assess chronic low-level inflammation.
Change in children's dietary habits | 2-weeks before intervention, during intervention (20 weeks), 2-weeks after intervention, and 2-weeks at 6 months follow-up
  Parents reported outcomes. Dietary habits are assessed via app diary (e.g. frequency and composition of meals).
Change in children's physical activity | 2-weeks before intervention, during intervention (20 weeks), 2-weeks after intervention, and 2-weeks at 6 months follow-up
  Parents reported outcomes. Physical activity is assessed via app diary (e.g., less sedentary time, increased physical activity).
Change in parent-reported quality of life in children | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Parents reported outcomes. Quality of Life is assessed with the KidScreen-27 questionnaire assessing the five dimensions physical well-being, psychological well-being, relationships with parents and autonomy, social support and peers and school environment. The KidScreen-27 consists of 27 items of which each is answered on 5-point Likert type scales with higher scores representing better quality of life

OTHER OUTCOMES:
Acceptance and usability of the app (parent reported outcome) | +22 weeks (Post intervention)
  The usability of the app is assessed using the eHealth App Usability Questionnaire (MAUQ). The questionnaire measures usability on three subscales (ease of use, Interface and satisfaction, usefulness). The MAUQ questionnaire consists of 18 items with a score ranging from 1 to 7. Score 7 means a better result.
Acceptance and usability of the app | During the intervention (20 weeks)
  The usability of the app is measured by means of how often and how long the parents use the app. The acceptance of the app is measured by means of dropout rate.
Exploratory: Metabolomic analysis of blood (biomarkers yet to be identified) | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Metabolomic analysis will be performed using the Nightingale Health's NMR-based metabolic biomarker profiling platform (https://research.nightingalehealth.com/biomarkers)
Exploratory: Proteomic analysis of blood (biomarkers yet to be identified) | Baseline, +22 weeks (Post intervention), +48 weeks (Follow-Up)
  Proteomic analysis will be performed using the Olink Target 96 Cardiovascular panels (https://olink.com/products-services/target/cardiometabolic-panel/)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias V. Kopp, Prof. Dr., Principal Investigator — Department of Paediatrics, Inselspital, Bern University Hospital, University of Bern, Switzerland; Michael Kaess, Prof. Dr., Principal Investigator — Universitäre Psychiatrische Dienste Bern (UPD), University of Bern, Switzerland
Locations (1):
- Department of Paediatrics, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch A, Wyssen A, Haupt C, Hammelbeck J, van Dorland HA, Fluck CE, Latzin P, Saner C, Jakob J, Kaess M, Kopp MV. Early Life Intervention in Paediatrics Supported by E-Health (ELIPSE)-a coaching app for parents to reduce obesity and second-hand smoke exposure in children: study protocols for two parallel-group randomised controlled trials. Trials. 2025 Nov 18;26(1):520. doi: 10.1186/s13063-025-09251-5. PMID 41254719